CLINICAL TRIAL: NCT01317550
Title: A Pilot Study of Minocycline and Armodafinil for Reducing the Symptom Burden Produced by Chemoradiation Treatment for Non Small Cell Lung Cancer
Brief Title: A Study for Reducing Symptom Burden Produced by Chemoradiation Treatment for Non Small Cell Lung Cancer by Minocycline and Armodafinil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2010-0872; R01 026582-26 (Other Grant/Funding Number: National Cancer Institute); NCI-2011-00778 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; Symptoms; Concurrent Chemoradiation; CXRT; Fatigue; Pain; Disturbed Sleep; Lack of Appetite; Drowsiness; Armodafinil; Nuvigil; Minocycline; Dynacin; Minocin; Minocin PAC; Myrac; Solodyn; Placebo
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Fatigue; Pain; Parasomnias; Anorexia; Sleepiness; cyclopia sequence | interventions — Modafinil; Sugars; Minocycline; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Armodafinil + Placebo (Experimental): Armodafinil orally 150 mg/day + Placebo capsules for 10 weeks
  Interventions: Drug: Armodafinil; Other: Placebo; Behavioral: Questionnaires
- Minocycline + Placebo (Experimental): Minocycline orally 100 mg twice/day + Placebo capsules for 10 weeks
  Interventions: Other: Placebo; Drug: Minocycline; Behavioral: Questionnaires
- Armodafinil + Minocycline (Experimental): Armodafinil orally 150 mg/day for 10 weeks + Minocycline orally 100 mg twice/day for 10 weeks
  Interventions: Drug: Armodafinil; Drug: Minocycline; Behavioral: Questionnaires
- Placebos (Placebo Comparator): Placebo Capsules orally once/day for 10 weeks
  Interventions: Other: Placebo; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Armodafinil — 150 mg by mouth once a day for a 10 week cycle.
  Other Names: Nuvigil
  Arms: Armodafinil + Minocycline; Armodafinil + Placebo
Other: Placebo — Capsules taken by mouth once a day for a 10 week cycle.
  Other Names: Sugar Pill
  Arms: Armodafinil + Placebo; Minocycline + Placebo; Placebos
Drug: Minocycline — 100 mg by mouth twice a day for a 10 week cycle.
  Other Names: Dynacin; Minocin; Minocin PAC; Myrac; Solodyn
  Arms: Armodafinil + Minocycline; Minocycline + Placebo
Behavioral: Questionnaires — Completion of symptom questionnaire before chemoradiation, then once a week during Weeks 1-16, takes up to 5 minutes to complete.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to compare armodafinil and minocycline when given alone or in combination to learn which is better for controlling symptoms, such as the side effects of chemoradiation, when given to treat lung cancer.

DETAILED DESCRIPTION:
The Study Drugs:

Armodafinil is designed to prevent excessive sleepiness.

Minocycline is an antibiotic. Minocycline has been shown to interrupt cytokine production, which may help to reduce multiple symptoms.

A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the roll of dice) to join 1 of 4 groups.

* Group 1 will take armodafinil and a placebo.
* Group 2 will take minocycline and a placebo.
* Group 3 will take armodafinil and minocycline.
* Group 4 will take placebos alone.

Neither you nor the study staff you will see in the clinic will know if you are receiving the study drug(s) and/or the placebo(s). However, if needed for your safety, the study staff will be able to find out which study drug you are receiving.

If needed, during this study, you may receive standard care by your treating doctors.

Study Drug Administration:

You will take the study drug(s)/placebos every day for 10 weeks. You should take the drug(s)/placebo(s) with a full glass of water. If you get an upset stomach, take them with food.

You will be given pamphlets with more information about how to take the study drugs/placebos.

You should bring your study drug/placebo capsules to the clinic every study visit.

Completing the Symptom Questionnaire:

Throughout the study, you will be asked to complete the symptom questionnaire. You will be asked about symptoms from therapy you may be experiencing and how they may be interfering with your daily activities. The study staff will either meet you during your regular clinic visit or call you at your home at a time that is convenient for you. In the clinic, you will complete the questionnaire by paper and pen, or by entering your answers into an electronic tablet computer. On the phone, study staff will ask you the questions and record your answers on paper or enter them into a computer. You will complete the symptom questionnaire before you begin chemoradiation and then 1 time a week during Weeks 1-16 of the study. The symptom questionnaire will take up to 5 minutes to complete.

Study Visits:

Before you begin chemoradiation:

* You will complete 4 questionnaires about pain and other symptoms, your mood, and your quality of life. Completing all 4 of the questionnaires will take about 15 minutes.
* If you are able to become pregnant, you will have a urine pregnancy test. The study staff will give you the pregnancy test kit at your scheduled visit, and will review and record the results of the test before you can pick up the study drugs from the pharmacy. The pregnancy test will be repeated at weeks 1, 4, 7, and 12 (or at the first follow-up clinic visit post-treatment) and 30 days after the study drugs are stopped .

During the last week of chemoradiation (about Week 7):

-You will complete 3 questionnaires about your symptoms, mood, and quality of life. These questionnaires will take about 10 minutes total to complete.

After about Week 7, the study staff will call you 1 time a week to check on you until Week 10. This phone call should last only a few minutes. If you have had several side effects from chemoradiation, this phone call may take longer.

About Week 12 (or at the first routine follow-up clinic visit post-treatment):

* You will complete the 3 questionnaires about your symptoms, mood, and quality of life.
* If you were smoking at the beginning of the study, you will complete a questionnaire that asks if you stopped smoking any time during the study. This will take a few minutes to complete.
* You will be asked to complete another questionnaire that asks about your satisfaction with the study drug(s). This will take a few minutes.

Length of Study:

You will be on study for about 16 weeks. You will take the study drug(s) for 10 weeks and complete the symptom survey until Week 16. You will be taken off study early if you have intolerable side effects.

This is an investigational study. Armodafinil is FDA approved and commercially available for the treatment of excessive sleepiness. Minocycline is FDA approved and commercially available for the treatment of bacterial infections. The use of these drugs to help reduce chemoradiation symptoms is investigational.

Up to 12 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a pathologically proven diagnosis of NSCLC and consented to concurrent chemoradiation therapy at MD Anderson.
2. Patients > or =18 years old
3. Patients who will receive chemoradiation with platinum/taxane-based chemotherapy and with a total radiation dose of > 50 Gy, per treating physician's assessment
4. Patients who speak English or Spanish (due to the novel research and its complexity, we are only accruing English or Spanish-speaking patients to the protocol)
5. Patients must be willing and able to review, understand, and provide written consent before starting therapy

Exclusion Criteria:

1. Patients who are taking medications or have conditions that potentially preclude use of any study medications or interventions, as determined by the treating physician
2. Patients who are enrolled in other symptom management or treatment clinical trials
3. Patients currently taking methylphenidate and/or dextroamphetamine.
4. Patients with a history of clinically significant cutaneous drug reaction, or a history of clinically significant hypersensitivity reaction, including multiple allergies or drug reaction as documented in the patient medical records
5. Patients with pre-existing psychosis or bipolar disorder.
6. Patients with pre-existing renal impairment: The screening cut off for serum creatinine >1.5 times upper limits of normal (ULN), according to MD Anderson testing standards, will be done by the oncologist to qualify for CXRT.
7. Patients with pre-existing hepatic impairment: The screening for total bilirubin >1.5 times ULN will be done by the oncologist to qualify for CXRT. The screening for > 2 times the upper limit of normal hepatotoxicity, alkaline phosphatase (ALP) and alanine aminotransferase (ALT) (and aspartate aminotransferase [AST] if it is ordered and available in the medical records) will be done by the oncologist to qualify for CXRT.
8. Patients with pre-existing Tourette's syndrome.
9. Patients with hypersensitivity to any tetracyclines.
10. Patients who are pregnant. Pregnancy will be confirmed by negative urine test. Study staff will provide the pregnancy kits to women and make sure the results are known and recorded in the follow-up notes in Clinic Station before additional study drug prescriptions are filled by the Pharmacy
11. Patients with uncontrolled cardiac disease, within the past six months history of left ventricular hypertrophy, myocardial infarction, and history of mitral valve prolapse syndrome with previous central nervous system (CNS) stimulant use.
12. Patients taking medicines that are strong CYP3A4 inhibitors or inducers (including conivaptan, indinavir, nelfinavir, ritonavir, nefazodone, and phenytoin), or strong CYP2C19 inhibitors (including citalopram and clopidogrel) .
13. Patients on vitamin K antagonist warfarin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhongxing Liao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.utmdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 15, 2011 to October 21, 2013. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Armodafinil: Armodafinil 150mg (capsule) once a day during entire course of radiation therapy for 10 weeks
- Minocycline: Minocycline 100mg (capsule) two times a day during the entire course of radiation therapy for 10 weeks
- Matching Placebo: Placebo capsules orally once/day for 10 weeks
Period: Overall Study
Arm/Group | Armodafinil | Minocycline | Armodafinil + Minocycline | Matching Placebo
Started | 5 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Lack of compliance study med | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Armodafinil+Minocycline: Armodafinil orally 150 mg/day for 10 weeks + Minocycline orally 100 mg twice/day for 10 weeks
- Total: Total of all reporting groups
Arm/Group | Armodafinil | Minocycline | Armodafinil+Minocycline | Matching Placebo | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 1 | 1 | 5
  >=65 years | 2 | 1 | 2 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.67 (7.09) | 60 (11.36) | 66.33 (8.08) | 65 (12.77) | 63.75 (8.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 2 | 6
  Male | 2 | 2 | 1 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 3 | 3 | 2 | 3 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Variable: Combined AUC of Selected Symptoms Fatigue, Pain, Disturbed Sleep, Lack of Appetite and Drowsiness
Description: Each item is rated on a 0 to 10 scale with 0 = symptom not present or no interference and 10 meaning the symptom severity is as bad as can be imagine or complete interference using the MD Anderson Symptom Inventory (MDASI). It is a measure of symptom burden, which includes symptom severity and how they interfere with daily functioning. For this study, the sub scale is the average of the 5 pre-selected items namely fatigue, pain, disturbed sleep, lack of appetite and drowsiness. This subscale ranges from 0 to 10. The primary outcome is the average of the 70-day area (10 week study) under the curve for the sub scale. AUC ranges from 0 (0*70) to 700 (10*70). To put this into perspective, the average AUC for the placebo group of 200.8 can also be thought of as 2.87 (200.8/70) on a 0 to 10 scale over the 70 day study period. Lower values represent better outcome. Higher values represent worse outcome.
Time Frame: During 10 weeks of CXRT
Population: Of the 14 randomized patients, 12 (85% were evaluable for the primary efficacy analysis).
Measure: Mean (Standard Deviation); unit: Units on a scale week
Groups:
- Armodafinil: Armodafinil 150mg (capsule) once a day during entire course of radiation therapy (10 weeks + 2 days
- Minocycline: Minocycline 100mg (capsule) two times a day during the entire course of radiation therapy (10 weeks + 2 days)
Arm/Group | Armodafinil | Minocycline | Armodafinil+Minocycline | Matching Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3
Units on a scale week
  Average AUC | 157.4 (181.4) | 81.1 (22.2) | 255.9 (65.3) | 200.8 (106.9)
  Fatigue | 259.3 (168.5) | 127.2 (60.5) | 372 (113.5) | 279.8 (193.6)
  Pain | 145.8 (233.6) | 114.5 (135.6) | 185.3 (121.) | 190 (96.7)
  Disturbed Sleep | 109.2 (165) | 80 (44.3) | 213.2 (81.5) | 224.7 (205.7)
  Lack of appetite | 133.3 (134.6) | 27.7 (28.1) | 298.3 (23.3) | 189 (72.6)
  Drowsiness | 139.3 (209.7) | 59.2 (32.8) | 210.7 (82.3) | 120.3 (69.5)

ADVERSE EVENTS:
Time Frame: Baseline up to 16 weeks
Description: All participants will be seen weekly in the radiation oncology clinics, allowing clinic and research staff to closely monitor potential adverse events during treatment. Participants will continue their symptom interventions for an additional 3 weeks after therapy is completed (when study treatment-related symptoms are at their peak)
Arm/Group | Armodafinil + Placebo | Minocycline + Placebo | Armodafinil + Minocycline | Placebos
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes